CLINICAL TRIAL: NCT06055959
Title: A Multicenter Open-Label, Uncontrolled Study to Evaluate the Pharmacokinetics, Pharmacodynamics, Safety, Tolerability, and Activity of Zilucoplan in Pediatric Study Participants From 2 to Less Than 18 Years of Age With Acetylcholine Receptor Antibody Positive Generalized Myasthenia Gravis
Brief Title: A Study to Evaluate Subcutaneous Zilucoplan in Pediatric Participants With Generalized Myasthenia Gravis
Acronym: ziMyG
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MG0014; U1111-1290-3349 (Other: World Health Organization (WHO)); 2022-502072-23 (Registry Identifier: EU Clinical Trials)
Record Dates: First submitted 2023-09-20; First posted 2023-09-28 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Generalized Myasthenia Gravis
Keywords: RA101495; gMG; generalized myasthenia gravis; zilucoplan; pediatric; MG0014
MeSH Terms: conditions — Myasthenia Gravis | interventions — zilucoplan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Zilucoplan Arm (Experimental): Study participants will receive zilucoplan in pre-defined dose based on their weight.
  Interventions: Drug: Zilucoplan

INTERVENTIONS:
Drug: Zilucoplan — Zilucoplan will be administered subcutaneously to pediatric study participants.
  Other Names: RA101495

SUMMARY:
The purpose of this study is to assess the pharmacokinetics, pharmacodynamics, safety, tolerability, immunogenicity and activity of zilucoplan (ZLP) in pediatric study participants with generalized myasthenia gravis (gMG).

ELIGIBILITY:
Inclusion Criteria:

United States of America (USA) specific inclusion criterion:

- Participant must be 12 to <18 years of age at the time of signing the Informed consent/assent according to local regulation

Rest of world (ROW) specific inclusion criterion:

- Participant must be 2 to <18 years of age at the time of signing the Informed consent/assent according to local regulation

Global inclusion criteria:

* Participant has a diagnosis of generalized myasthenia gravis (gMG) confirmed by a prior positive serologic test result to acetylcholine receptor (AChR) prior to Screening
* Participant meets the criteria as defined by the Myasthenia Gravis Foundation of America (MGFA) Clinical Classification II to IV at Screening
* Participants with gMG, including:
* An MG-activities of daily living (MG-ADL) total score of 6 or more in adolescents from 12 years to <18 years of age at Screening
* Documented weakness in at least 1 limb, neck, or bulbar muscle in children from 2 years to <12 years of age at Screening (does not apply to US)
* Documented vaccination against meningococcal infections within 3 years prior to study start. If not fully vaccinated, participants must receive appropriate prophylactic antibiotic treatment until at least 2 weeks after the initial dose of vaccine(s)

Exclusion Criteria:

* Participant has known positive serology for muscle-specific kinase
* Participant has any medical or psychiatric condition that, in the opinion of the Investigator, could jeopardize or would compromise the participant's ability to participate in this study
* Participant has had a thymectomy within 6 months prior to Baseline
* Participant has minimal Manifestation Status of MG based on the clinical judgement of the Investigator
* Current or recent systemic infection within 2 weeks prior to Baseline or infection requiring intravenous antibiotics within 4 weeks prior to Baseline

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Estimated)
Dates: Start 2024-10-16 (Actual); Primary Completion 2026-11-16 (Estimated); Study Completion 2026-12-25 (Estimated)

PRIMARY OUTCOMES:
Plasma concentrations of zilucoplan (ZLP) sampled at Week 4 (Day 29) | Week 4 (Day 29)
  Blood samples will be collected for measurement of plasma concentrations of ZLP on Day 29 predose.
Change from Baseline in sheep red blood cell (sRBC) lysis at Week 4 (Day 29) | Week 4 (Day 29)
  Samples for measurement of sRBC lysis will be collected on Day 29 predose.
Change from Baseline in complement component 5 (C5) levels at Week 4 (Day 29) | Week 4 (Day 29)
  Samples for measurement of C5 will be collected on Day 29 predose.

SECONDARY OUTCOMES:
Occurence of treatment-emergent adverse events (TEAEs) during the course of the study | From Baseline (Day 1) to Safety-Follow-Up Visit (up to Week 15)
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Occurrence of treatment-emergent serious adverse events (TESAEs) | From Baseline (Day 1) to Safety-Follow-Up Visit (up to Week 15)
  A serious adverse event (SAE) is defined as any untoward medical occurrence that, at any dose:
  Results in death Is life-threatening Requires inpatient hospitalization or prolongation of existing hospitalization Results in persistent disability/incapacity Is a congenital anomaly/birth defect Important medical events
Occurrence of TEAEs leading to permanent withdrawal of investigational medicinal product (IMP) | From Baseline (Day 1) to Safety-Follow-Up Visit (up to Week 15)
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. AEs leading to permanent withdrawal of study medication.
Occurrence of treatment-emergent infections | From Baseline (Day 1) to Safety-Follow-Up Visit (up to Week 15)
  Percentage of participants who experienced treatment-emergent infections as adverse events.
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment.
Occurrence of antidrug antibody (ADA) and anti- polyethylene glycol (PEG) antibodies at Week 4 (Day 29) | Week 4 (Day 29)
  ADA and anti-PEG antibodies will be evaluated in serum samples.
Change in MG-activities of daily living (MG-ADL) score from Baseline to Week 4 (Day 29). | Week 4 (Day 29)
  The MG-ADL score is an 8-item patient-reported outcome (PRO) instrument. The MG-ADL targets symptoms and disability across ocular, bulbar, respiratory, and axial symptoms. The item responses are scored from 0 to 3, and the total score of MG-ADL is the sum of the 8 items and ranges from 0 to 24, with a higher score indicating more disability.
Change in Quantitative MG (QMG) score from Baseline to Week 4 (Day 29) | Week 4 (Day 29)
  QMG score is a standardized and validated quantitative strength scoring system that was developed specifically for MG. The QMG total score is obtained by summing the responses to each individual item (13 items; Responses: None=0, Mild=1, Moderate=2, Severe=3). The score ranges from 0 to 39, with lower scores indicating lower disease activity.
Myasthenia Gravis Foundation of America Post-Interventional Status (MGFA-PIS) at Week 4 (Day 29) | Week 4 (Day 29)
  The MGFA-PIS is a physician-determined assessment of clinical symptoms of MG after initiation of MG specific therapy. For the purpose of the current study, Minimal Manifestation will be determined at each scheduled time point after treatment initiation (rather than after 1 year). Change in status (improved, unchanged, worse, exacerbation, or died of MG) will also be determined.
Change in Pediatric Quality of Life Inventory (PedsQoL), Version 4 domain scores from Baseline to Week 4 (Day 29) | Week 4 (Day 29)
  The PedsQoL generic core scale (Version 4) is a validated instrument that is suitable for use with pediatric populations. PedsQoL generic core scales assess Physical Functioning, Emotional Functioning, Social Functioning, and School Functioning. The scale has 23 items with a score range of 0 to 4. Following transformation, the score range of each domain as well as the total score is 0-100 with higher scores indicating higher HRQoL.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (9):
- United States (2):
  - Mg0014 50168, Chicago, Illinois
  - Mg0014 50574, Denton, Texas
- Mg0014 40144, Milan, Italy
- Poland (2):
  - Mg0014 40774, Katowice
  - Mg0014 40218, Warsaw
- South Korea (2):
  - Mg0014 20104, Seoul
  - Mg0014 20220, Seoul
- United Kingdom (2):
  - Mg0014 40735, Glasgow
  - Mg0014 40736, London

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this study may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed.All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: http://www.Vivli.org